CLINICAL TRIAL: NCT00890578
Title: It is Our Intent to Conduct a Prospective Randomized Controlled Trial Examining the Use of Histoacryl© in the Closure of Surgical Incisions in Comparison to Subcuticular Suture and to Dermabond©.
Brief Title: HISTOACRYL: A Study of Its Efficacy in Final Scar Formation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Galen Perdikis, M.D., Mayo Clinic
Other Study IDs: 08-007642
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Surgical Incisions
Keywords: Histoacryl; closure of surgical incisions
MeSH Terms: conditions — Surgical Wound | interventions — octyl 2-cyanoacrylate; Enbucrilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1-abdominal: half abdominal surgeries (20 patients out of 40)
  Interventions: Procedure: adhesive to suture
- 2-breast: half breast surgeries (20 out of 40)
  Interventions: Procedure: adhesive to suture

INTERVENTIONS:
Procedure: adhesive to suture — surgical closure
  Other Names: Dermabond, Histoacryl, or sutures --patients could be randomized to.

SUMMARY:
The use of tissue adhesives for the closure of surgical incisions is becoming increasingly common. Several publications exist purporting the equivalence of tissue adhesive to suture with regard to dehiscence, infection, and cosmesis. Two of the most frequently used adhesives are Histoacryl© and Dermabond©. Despite their popularity, only one study exists comparing the two. In this non-English study only small wounds in an exclusively pediatric population were studied (12). Operative time, cost, and objective measures of scar size were not examined. In the present study we aim to evaluate the relatively large surgical incisions resulting from breast reduction, mastopexy, panniculectomy, and abdominoplasty closed with either Histoacryl©, Dermabond©, or subcuticular suture. The primary aim is to investigate differences in time to wound closure. Secondary aims are to compare the three approaches with respect to cost, dehiscence, infection, scar size, and cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* Age: Younger than 21
* Gender: Females only. Given the nature of the procedures, as well as our clinical experience, we cannot anticipate recruiting enough male patients to be able to evaluate them as a subgroup. Since there may be differences in distributions of measures, to keep the groups more homogeneous we plan to recruit only females from the outset. Having either:
* Reduction Mammoplasty or mastopexy patients:

  * Patients who present to the plastic surgery clinic and are scheduled for breast procedures will be recruited and consented by a clinical studies co-ordinator.
  * This will include patients undergoing a standard Wise pattern reduction mammoplasty (reduction and lift) or a standard Wise pattern mastopexy (lift only). See exclusion criteria below.
* Abdominoplasty or panniculectomy patients:

  * Patients who present to the plastic surgery clinic and are scheduled for abdominal procedures will be recruited and consented by a clinical studies coordinator. See exclusion criteria below.

Exclusion Criteria:

* Though women of childbearing age will be allowed to participate in this study, no pregnant patients will be enrolled.
* Patients with any factors that may have an adverse effect on wound healing:

  * previous hypertrophic scars or keloid
  * known vitamin C deficiency
  * known zinc deficiency
  * smoking
  * steroid use
  * known connective tissue disorder
  * hypoalbuminemia
  * any factor not listed that the attending consultant seeing the patient feels would adversely effect wound healing.
* Patients who have a known sensitivity to adhesives

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1) and 2): Reduction Mammoplasty or mastopexy patients: Patients who present to the plastic surgery clinic and are scheduled for breast procedures will be recruited and consented by a clinical studies co-ordinator. This will include patients undergoing a standard Wise pattern reduction mammoplasty (reduction and lift) or a standard Wise pattern mastopexy (lift only). See exclusion criteria below.
  1) and 2): Abdominoplasty or panniculectomy patients: Patients who present to the plastic surgery clinic and are scheduled for abdominal procedures will be recruited and consented by a clinical studies coordinator. See exclusion criteria below.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Histoacryl© to Dermabond© is lacking. Investigation of Histoacryl© in direct comparison to Dermabond© as well as to suture. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Galen Perdikis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States